CLINICAL TRIAL: NCT04748731
Title: Internet Mentalization-based Video Feedback Intervention to Improve Parental Sensitivity in Mother-infant Dyads With Maternal Depressive Symptoms: Randomized Controlled Feasibility Trial
Brief Title: Video Feedback to Improve Parental Sensitivity in Mother-infant Dyads With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Instituto Milenio para Investigación en Depresión y Personalidad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VF and mentalizing
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2021-01

CONDITIONS: Parent-Child Relations; Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group. Video-feedback intervention. (Experimental): A weekly online brief intervention using video-feedback and psycho-educational materials on early parenting (detailed description of the intervention on section 5).
  Interventions: Behavioral: Internet mentalization-based video feedback intervention to improve parental sensitivity in mother-infant dyads with maternal depressive symptoms
- Control Group. Psycho-educational intervention (Other): They will receive weekly information on parenting in the 1st year of life. They will have direct contact (via WhatsApp) with a child psychologist to ask questions about the material and to refer to specialized support if needed.
  Interventions: Behavioral: Psycho-Educational Intervention

INTERVENTIONS:
Behavioral: Internet mentalization-based video feedback intervention to improve parental sensitivity in mother-infant dyads with maternal depressive symptoms — a weekly online brief intervention using video-feedback and psycho-educational materials on early parenting
  Arms: Experimental Group. Video-feedback intervention.
Behavioral: Psycho-Educational Intervention — Reception of psycho-educational materials
  Arms: Control Group. Psycho-educational intervention

SUMMARY:
Title: "Internet mentalization-based video feedback intervention to improve parental sensitivity in mother-infant dyads with maternal depressive symptoms: randomized controlled feasibility trial". Funding: ANID Millennium Science Initiative /Millennium Institute for Research on Depression and Personality-MIDAP ICS13_005 (MIDAP, www.midap.org).

Principal Investigator: Marcia Olhaberry Huber, PhD, Academic, School of Psychology, Pontificia Universidad Católica de Chile, Associate Researcher, MIDAP.

MIDAP Research Team: Javier Moran, PhD. Academic at the University of Valparaíso, María José León, PhD, Stefanella Costa, PhD. and Fanny Leyton, PhD. (c) University of Valparaíso.

General Objective: To evaluate feasibility and acceptability of a brief Internet mentalization-based video feedback intervention to improve sensitivity in mothers with depressive symptoms. Key parameters for a future effectiveness study will be identified

Design: Pilot randomized clinical trial; Participants: 60 mother-infant dyads (aged 4-12 months) attended in Public Health Centres.30 dyads will be assigned to the experimental group (EG) and will receive a weekly online brief intervention using video-feedback and psycho-educational materials on early parenting. 30 dyads will be assigned to the control group (CG) and will receive only psycho-educational materials. The study includes 3 assessments (pre-intervention, post-intervention and follow-up) and four weekly intervention sessions. Data analysis: For quantitative data descriptive statistics and ANCOVA will be used, for qualitative data Grounded Theory.

DETAILED DESCRIPTION:
Background A growing body of research recognises the key role of both parental sensitivity and mentalizing in fostering positive parent-child relationships. This, in turn, is fundamental for a child's mental health and intergenerational transmission of attachment.

Parental sensitivity concerns a parent's ability to perceive and interpret their child's cues accurately and to respond accordingly in a contingent manner (Ainsworth et al., 1978). Parental sensitivity has been associated with the development of attachment and general socio-emotional development in childhood. The association between parental sensitivity and cognitive variables like joint attention, executive functioning development in early childhood and Theory of Mind in preschoolers has also demonstrated it.

The caregiver's capacity to think of his/her child in terms of mental state (i.e., parental mentalizing or parental reflective functioning) is linked with the development of affect regulation in the child, with the intergenerational transmission of attachment and with the development of social and reflective abilities in childhood. Evidence also suggests that mentalizing may constitute a protective factor for the transmission of psychopathology in childhood.

*THE INTERVENTION*

The present intervention aims to improve parental sensitivity and mentalizing in depressed mothers using a model based on video-feedback methodology in an online modality.

The whole intervention consists of 4 sessions plus 1 pre-intervention assessment session. Additionally, there is 1 weekly group supervision, along with the therapist independent work on the case between sessions. Each intervention's session has the same structure: Checking outcomes from the previous session; Videofeedback; New video recording; Post-interview; Tasks definition.

Between each session, the therapist analyses the material independently and attends group supervision. Each element of the intervention is described in detail below.

PRE-INTERVENTION ASSESSMENT Methodology: Online, delivered by a trained clinical psychologist Duration and frequency: 90 minutes, once.

1. Questionnaires and scales:

   1. Sociodemographic information questionnaire
   2. Children social-emotional screening (ASQ SE).
   3. Mothers depressive symptoms (Edinburgh Postnatal Depression Scale; EDPS; Patient Health Questionnaire; PHQ-9)
2. Video recording of free mother-baby play at the end of the session (coded with the Emotional Availability Scale; EAS).
3. MINI PDI interview (after video recording).
4. Childhood Trauma Questionnaire Short Form (CTQ-SF)
5. Examination of the mother's concerns regarding the child, their relationship, or her as a mother. Discussion of the mother's reason for referral and intervention goals definition, integrating the mother's concerns.

THERAPIST INDEPENDENT WORK General Description: Review of case's background information, video analysis and VF script elaboration Duration and frequency: 60 minutes weekly. The free play video -recorded in the initial assessment is watched and analysed, and then resources and opportunities are identified.

The intervention's goal is defined considering the mother's concerns and the reason for referral defined in the initial assessment.

Segments of 30 and 60 seconds are selected by stopping the video at the end of the interaction sequence. Both the start and end's times are written down on the script. It is recommended to show the complete video unless negative segments are identified (i.e., segments in which the mother appears as hostile or insensitive when the child appears severely under-regulated). In such cases, it might be necessary to consider only the positive sequences or selecting specific images within the video.

Specific goals to be achieved in each selected segment must be identified. Comments and questions to be made by the therapist should be defined, and these should be linked to each selected segment's goal.

SUPERVISION Methodology: Online group supervision. Duration and frequency: 120 minutes weekly. Guidelines: Two guidelines are provided and examined. These documents were developed to orient both online psychotherapeutic processes in early childhood and psychotherapeutic interventions using video feedback in 0-5 years old children.

After the therapist prepares their first case, they must present to the group at least 1 complete VF process. Then, they must present parts of the other cases they will address. In the first case, the therapist must present a comprehensive diagnosis of the case integrating the initial assessment results, the complete videos, the completed analyses, the segment selected and the elaborated script. At further sessions, the therapist would have to present not the whole process but only particular aspects of each case or about his work as a therapist.

The supervision has a reflective methodology, and the experience of each of the intervention's participants is considered (i.e., supervisor, child, caregiver and therapist). In the supervision space, the supervisor can also act as a supportive figure for the therapist.

INTERVENTION'S SESSIONS Methodology: Online and delivered by the same therapist that made the initial assessment. Duration and frequency: 60 minutes weekly.

Checking outcomes from the previous sessions. Starting from session 2. A space for discussing the caregiver's perceptions about changes in the relationship related to the former session's tasks.

Video Feedback. The topic of each session addresses the contents of the video recorded in the previous session. First, the structure of the session is explained to the mother. Next, the mother is asked about the video recorded -this is useful to check if what she remembers is consistent with what was observed-. After that, the Video Feedback intervention's goal is presented to the mother, explaining its benefits and exploring their perceptions around this issue.

Then, the video sequences previously selected are shown. Before commenting, it is important to ask the mother to observe and describe objectively (i.e., without making inferences) what she is watching, to check that both caregiver and therapist are watching the same and therefore, reflecting about the same contents. For example, a caregiver watching a video might say "my son does not want to play with me" when the child is focused on playing with a toy. In those cases, it can be useful to ask the mother again to describe what was watched without interpreting. In this way, we check that we are both watching the same, which is key for our comments to be well received.

Video Recording. Each session has a moment when a new interaction following a new instruction is recorded (e.g., playing, feeding, singing).

Post-Interview. After each video recording, a semi-structured interview is carried out with the following questions:

(About the mother herself) What was the most pleasant aspect of the interaction with your baby? Why? What was the most difficult aspect of the interaction with your baby? Why? (About the baby) What do you think was the most pleasant aspect of the interaction for your baby? What made you think that ___ was the most pleasant aspect for your baby? What do you think was the most difficult aspect of the interaction for him/her? What made you think that___ was the most difficult aspect for him/her? (About the interaction) Has this type of interaction with your baby happened before? (if yes) Could you please give me an example? Could you describe what caught your attention or what you learned about yourself, your baby or your relationship after this interaction?

Tasks definition: behaviours or activities to perform during the week are defined. These can be proposed by the therapist or emerge from what the mother learnt in the video feedback. Examples: playing 5 minutes, 3 times per week with; observe the baby's preferences in a specific context, support the baby in reaching a new ability; among others.

*THE STUDY*

Design: Cluster randomized controlled trial feasibility and pilot study

Participants: Mothers presenting depressive symptoms will be invited from three public primary health centres from Santiago, Valparaíso and Puerto Varas. Sample size will be 60 (control group [CG]=30; experimental group [EG]=30), based on similar studies and general recommendation for pilot studies1819.

Professionals delivering the intervention must be psychologists with at least 1 year of experience.

Procedure: Participants will be invited by a primary health worker. On participation agreement, they will be contacted to perform the first interview to assess eligibility and sign an informed consent (as established by the PUC Ethical Committee). After that, participants will be randomized to CG or EG in a 1:1 ratio. A random number sequence will be computer-generated in varying block sizes (2&4) and stratified by centre.

Based on a mentalization-based VFI developed by Olhaberry and colleagues aimed to improve maternal sensitivity, a 4 sessions internet VFI will be manualized. Therapists will be trained in the model over 3 days (24 hours) and then supervised session by session. The CORE-OM and an assessment of the therapist's adherence to the model will be used during supervision. For this purpose, each session will be video recorded.

CG, psycho-educational intervention: They will receive weekly information on parenting in the 1st year of life. They will have direct contact (via WhatsApp) with a child psychologist to ask questions about the material and to refer to specialized support if needed.

Outcome measures will be taken before the first session, after treatment, and in a 3 -months follow up period.

Instruments: 1. Sociodemographic information questionnaire; Parental Sensitivity (Primary Outcome; Emotional Availability Scale; EAS; 2. Secondary outcomes: Parental Reflective Functioning (Parent Development Interview-Revised, Short Version; PDI-R); Children Social-emotional screening 3. Covariates: Mothers depressive symptoms (Edinburgh Postnatal Depression Scale; EDPS; Patient Health Questionnaire; PHQ-9); Childhood Trauma Questionnaire Short Form (CTQ-SF)

Analysis plan

Quantitative Outcomes: Descriptive statistics to establish CG's and EG's clinical and sociodemographic variables, eligibility and recruitment rate, and adherence. ANCOVA will be used to determine differences between groups, controlling for a baseline for each outcome.

Observational measures will be applied by a certified pair of coders. Cohen-kappa will be used for Inter-rater reliability. Qualitative study: to assess participant's satisfaction with the intervention, semi-structured interviews will be conducted after the trial's end. 4 mothers from each centre will be interviewed, selected according to the presence/absence of change in the main outcome (2 presenting change/2 not presenting change, to ensure variability). Additionally, a focus group will be performed with VF therapists (3 professionals for each centre; 9 in total). Interviews aim to collect information regarding the feasibility of performing the intervention and also training and supervision experience. Interviews' data will be analyzed using Grounded Theory´s open coding.

ELIGIBILITY:
Inclusion Criteria:

* Mother must be over 18 years old
* Mother must have a 4 to 12 months infant
* Mother must be a user of primary public health
* Mother must score at least 5 points in the EPDS during routine health controls in health centres

Exclusion Criteria:

* Mothers presenting severe intellectual deficit or psychotic symptoms.
* Infants presenting developmental disorders and/or at high risk of abuse or neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Change in Maternal sensitivity | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  Emotional Availability Scale (EAS). Scores range from 0 to 10o with higher scores indicating higher emotional availability. Therefore, higher scores mean better outcomes.

SECONDARY OUTCOMES:
Change in Parental Reflective Functioning | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  Reflective Functioning Scale. Scores range from 0 to 10 with higher scores indicating higher reflective functioning, therefore, higher scores mean better outcomes.
Change in Maternal Depressive Symptoms Measured with EPDS | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  Edinburgh Postnatal Depression Scale (EPDS). Scores range from 0 to 30 with higher scores meaning higher depressive symptomatology. Therefore, higher scores mean worst outcomes.
Change in Maternal Depressive Symptoms Measured with CORE OM | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  CORE OM. Scores range from 0 to 136 with higher scores meaning higher depressive symptomatology. Therefore, higher scores mean worst outcomes.
Change in Maternal Depressive Symptoms Measured with PHQ 9 | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  Patient Health Questionnaire (PHQ-9). Scores range from 0 to 27 with higher scores meaning higher depressive symptomatology. Therefore, higher scores mean worst outcomes.
Change in Children Socio Emotional Development | before the intervention; through study completion, an average of 1 year; and a 3 months follow-up.
  Ages and Stages Questionnaire (ASQ-SE). Scores range from 0 to 75 with higher scores meaning lower socio-emotional development. Therefore, higher scores mean worst outcomes.

OTHER OUTCOMES:
Feasibility of the intervention | Through study completion, approximately 18 months
  Estimate the proportion of performed sessions versus planned sessions and number of participants who remain in the study during intervention and follow up period. Higher scores mean better outcomes.
Intervention's acceptability by credibility/expectancy rates | Through study completion, approximately 18 months
  Credibility/Expectancy Questionnaire (CEQ).Scores range from 0 to 100 with higher scores indicating higher acceptability of the intervention. Therefore, higher scores mean better outcomes.
Intervention's acceptability by participant's experience | Through study completion, approximately 18 months
  In-Depth interview to explore the participant's experience

CONTACTS AND LOCATIONS:
Locations (1):
- CESFAM Puerto Varas, Puerto Varas, Los Lagos Region, Chile

REFERENCES:
- [Derived] Olhaberry M, Leyton F, Moran-Kneer J, Leon MJ, Sieverson C, Muzard A, Honorato C, Ensink K, Malberg N, Luyten P, Costa-Cordella S. Strength-based Video-feedback to improve maternal sensitivity in mother-infant dyads with maternal depressive symptoms: Study protocol for a randomized controlled feasibility trial. Medwave. 2022 Dec 15;22(11):e2570. doi: 10.5867/medwave.2022.11.2570. English, Spanish. PMID 36583684